CLINICAL TRIAL: NCT02673996
Title: The Pathophysiological Role of Adrenergic Antibodies in Postural Tachycardia Syndrome (Aims #1&2)
Brief Title: POTS Adrenergic Ab (CIHR Aims #1&2)
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Satish Raj, Professor, University of Calgary
Other Study IDs: REB15-2434; MOP142426 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postural Tachycardia Syndrome
Keywords: antibody; autoimmune; adrenergic; autonomic
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Phenylephrine; Isoproterenol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum for antibody assay; plasma for cytokine assessment; plasma for catecholamines
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Postural Tachycardia Syndrome (POTS): Patients with postural tachycardia syndrome; patients will receive both IV phenylephrine and IV isoproterenol
  Interventions: Drug: Phenylephrine; Drug: Isoproterenol
- Healthy (control) Subjects: Healthy volunteers that are gender and age-matched (by groups) to the POTS patients; healthy subjects will receive both IV phenylephrine and IV isoproterenol
  Interventions: Drug: Phenylephrine; Drug: Isoproterenol

INTERVENTIONS:
Drug: Phenylephrine — incremental small doses of IV phenylephrine to find the dose that transiently raises systolic blood pressure by 25 mmHg
  Other Names: NeoSynephrine
Drug: Isoproterenol — incremental small doses of IV isoproterenol to find the dose that transiently raises heart rate by 25 bpm
  Other Names: Isuprel

SUMMARY:
Objective: In this pilot study, we will test the hypothesis that patients with POTS (age 18-60 years) will have a higher percentage of functional antibodies to adrenergic receptors compared with control subjects without POTS.

DETAILED DESCRIPTION:
Background & Rationale:

Postural Tachycardia Syndrome (POTS) is a chronic state of orthostatic tachycardia (> 30 bpm increment from lying to standing) and typical symptoms that are worse on standing, and are relieved by lying down. Typical orthostatic symptoms include palpitation, lightheadedness, chest pains, dyspnea, tremulousness, blurred vision and mental clouding. POTS often occurs in younger individuals with a female predominance (4-5 fold). Using the RAND36 quality of life (QOL) tool, we showed that POTS patients had lower quality of life (QOL) scores than healthy subjects for both physical (26±9 vs. 54±6; P<0.0001) and mental health domains (43±11 vs. 52±10; P<0.0001). These QOL scores are similar to scores for chronic obstructive pulmonary disease and congestive heart failure.

In collaboration with the Kem/Yu lab (Oklahoma University), the investigators sought to determine whether POTS patients had functionally significant adrenergic receptor (AR) Abs. Samples from 14 POTS patients (included 7 blinded, well-characterized samples from Vanderbilt) and 10 healthy control subjects. Using the rat cremaster artery assay, the sera/immunoglobulin (IgG) of the POTS patients demonstrated significantly greater arteriolar contractile activity (69±3% of baseline vessel diameter) compared to the control subjects (91±1% of baseline; P<0.001). This contractility was suppressed with prazosin, an α1-AR blocker. With the addition of POTS sera, the phenylephrine dose-response curve was shifted to the right. In other words, a higher dose of phenylephrine was required to achieve the same degree of vasoconstriction, suggests that the α1-AR Ab is actually a partial-agonist/antagonist.

Using a cell-based cyclic AMP (cAMP) reporter assay, all POTS sera had dose-dependent β1-AR activation (max: +30±3% from buffer baseline) compared to control sera (-1±2% from buffer baseline; P<0.001), and 7/14 POTS patients (but no control subjects) had elevated β2-AR activation. The excessive β1-AR activation could be blocked with propranolol. With the addition of POTS sera, the isoproterenol dose-response curve was shifted to the left (a lower isoproterenol dose was required to achieve the same receptor activation in the presence of the POTS sera). These data suggest that the β1-AR Ab is actually a straight agonist.

Big Picture:

While exciting, these data are obtained from only 14 POTS patients. In this protocol (Aim#1; REB15-2434), the investigators will study a larger cohort of POTS patients and control subjects in order to have a better sense of the true prevalence of these antibodies, to determine their association with other autoimmune illnesses, and to see if they relate to the patient-reported onset of illness.

In addition to this, the investigators seek to see whether this is physiologically significant in intact humans in vivo (Aim#2).

The investigators propose to perform dose response studies for phenylephrine and isoproterenol in POTS patients and control subjects with blood pressure (BP) and heart rate (HR) as the output metric and will then determine if these are different between POTS patients and control subjects and, more importantly, based on the auto-antibody in vitro activity.

Specifically, the investigators will give a series of injections of small doses of phenylephrine while monitoring their HR and continuous BP. After each injection, the investigators will note the peak BP increase and will monitor the patient until the BP returns to baseline. The investigators will give incrementally larger doses until the endpoint is achieved. The endpoint is the lowest test dose of phenylephrine that will increase the systolic BP by >25 mmHg (PHE-PD25).

the investigators will then repeat the same process with small doses of isoproterenol with the same monitoring. After each injection, the investigators will note the peak HR increase and will monitor the patient until the HR returns to baseline. The investigators will give incrementally larger doses until the endpoint is achieved. The endpoint is the lowest test dose of isoproterenol that will increase the HR by >25 bpm (ISO-PD25).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been previously diagnosed with POTS
* Control subjects (patients not diagnosed with POTS)
* Age between 18 - 60 years
* Males and Females (Give that >80% of POTS patients are female, we will attempt to enroll a similar percentage of female control subjects)
* Able and willing to provide consent

Exclusion Criteria:

* Smokers
* Overt cause for postural tachycardia, i.e., acute dehydration
* Significant cardiovascular, pulmonary, hepatic, or hematological disease by history or prior testing
* Highly trained athletes
* Subjects with somatization or severe anxiety symptoms will be excluded
* Use of drospirenone (a spironolactone analogue) containing oral contraceptive agent
* Hypertension defined as supine resting BP>145/95 mmHg off medications or needing antihypertensive medication
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule
* Unable to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with POstural Tachycardia Syndrome (POTS)
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of alpha-1 Ab titer positive subjects | 1 Year (to measure Adrenergic antibody assay)
  The primary comparison will be the proportion of Ab titers between POTS patients compared to control subjects.

SECONDARY OUTCOMES:
Antibody Positivity by Joint Hypermobility Status | 1 Year (to measure Adrenergic antibody assay)
  These comparisons include proportions of POTS patients with +va adrenergic Ab with a co-diagnosis of joint hypermobility syndrome (EDS III) vs without joint hypermobility syndrome (EDS III).
Antibody Positivity by Clinical Autoimmune Syndromes | 1 Year (to measure Adrenergic antibody assay)
  These comparisons include proportions of POTS patients with +ve adrenergic Ab with a co-diagnosis of a clinical autoimmune disorder vs without a clinical autoimmune disorder.
Antibody Positivity by Viral Onset of POTS | 1 Year (to measure Adrenergic Antibody assay)
  These comparisons include proportions of POTS patients with +ve adrenergic Ab with a viral onset to their POTS vs without a viral onset to their POTS.
Isoproterenol HR Increase (PD25) | 1 Year (to measure Adrenergic Antibody assay)
  A comparison of the dose of isoproterenol required to acutely increase the Heart Rate by 25 bpm from a pre-injection baseline (as a measure of beta-receptor sensitivity) in antibody positive vs. antibody negative subjects.
Phenylephrine Systolic BP Increase (PD25) | 1 Year (to measure Adrenergic Antibody assay)
  A comparison of the dose of phenylephrine required to acutely increase the Systolic Blood Pressure by 25 mmHg from a pre-injection baseline (as a measure of alpha-receptor sensitivity) in antibody positive vs. antibody negative subjects.
The proportion of beta adrenergic Ab titer positive subjects | 1 Year (to measure Adrenergic Antibody assay)
  The primary comparison will be the proportion of Ab titers between POTS patients

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No